CLINICAL TRIAL: NCT04635072
Title: Is 100% Pure Stabilized Whole Rice Bran (SWRB) Effective When Used as a Cleanser and an Emollient in Patients With Mild to Moderate Atopic Dermatitis?
Brief Title: Stabilized Whole Rice Bran (SWRB) for Mild to Moderate Atopic Dermatitis
Acronym: SWRB
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: RCSI & UCD Malaysia Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC 50
Record Dates: First submitted 2020-11-04; First posted 2020-11-18 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Patients with mild AD will be given SWRB in powder form, to be used as a cleanser after adding water to it according to set proportions given as instructions, one time per day.
  Patients with moderate disease will be instructed to use SWRB as a cleanser as above. In addition, they will also use SWRB as an emollient after constituting it into a paste as in instructions, apply at night and leave it overnight.
  The patients will be followed up for four to six weeks and the clinical features tabulated. Where appropriate, photographs of the lesion/s will be taken for evaluation of progression / regression at the end of the study, while protecting the identity of the patient.
  A questionnaire using the Likert scale, will be prepared for the patient's parent/s to complete. This will be to assess:
  * Parents' opinion of the product
  * Ease of application
  * Convenience (cleaning the bed of the powder, etc.)
  * Parents' perception regarding improvement seen/not seen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stabilised Whole Rice Bran (SWRB) (Experimental): Patients with mild AD will be given SWRB in powder form, to be used as a cleanser after adding water to it according to set proportions given as instructions, one time per day.
  Patients with moderate disease will be instructed to use SWRB as a cleanser as above. In addition, they will also use SWRB as an emollient after constituting it into a paste as in instructions, apply at night and leave it overnight.
  Interventions: Drug: Stabilised Whole Rice Bran

INTERVENTIONS:
Drug: Stabilised Whole Rice Bran — Patients with mild Atopic Dermatitis (AD) will be given SWRB in powder form, to be used as a cleanser after adding water to it according to set proportions given as instructions, once a day. Patients with moderate disease will use SWRB as a cleanser. In addition, they will also use SWRB as an emollient.
  Other Names: SWRB

SUMMARY:
This clinical trial serves to look at the effectiveness of SWRB for the treatment of mild to moderate Atopic Dermatitis in patients below the age of 18. Atopic Dermatitis (AD) is a common condition seen in dermatology, paediatric and primary care clinics in Malaysia. AD poses a significant biopsychosocial burden among sufferers and their families. Current management patterns of AD sufferers in South-east Asia mainly involve use of topical moisturizers and topical corticosteroids.

Rice bran and products derived from it have been studied regarding their anti-oxidant, nutritional, cholesterol lowering and health promoting properties. However, there are very few studies that have focused on the benefits of SWRB when used topically.

SWRB is cost-effective and easily available, while being an under-utilised product. The investigators wanted to study its effectiveness in controlling the signs and symptoms of Atopic Dermatitis when used as a cleanser and topical paste (emollient) as very little is known on this subject.

The investigators wish to study participants below 18 years of age with mild and moderate Atopic Dermatitis.

The participants will be followed up for four to six (4 - 6) weeks and the clinical features tabulated. This study does not involve any enteral or parenteral administration of SWRB.

Neither does it involve any invasive procedures.

DETAILED DESCRIPTION:
Objective of the study To study whether the natural product, SWRB, is effective to control the symptoms and signs of mild to moderate Atopic Dermatitis (AD)

Background, rationale & justification.

1. Atopic Dermatitis is a common condition seen in dermatology, paediatric and primary care clinics in Malaysia. The overall prevalence of Atopic Dermatitis in the paediatric population in Malaysia was shown to be around 13.4% in 2018 (Goh et al., 2018)
2. AD poses a significant biopsychosocial burden among sufferers and their families. (Carroll et al., 2005). Current management patterns of AD sufferers in South-east Asia mainly involve use of topical moisturizers and topical corticosteroids (Chan et al., 2006).
3. There are many concerns among parents of sufferers of AD regarding the side effects of these therapies, causing them to seek alternative therapies (Lee and Bielory, 2010).
4. Many emollients are available in the market which are either occlusives, hemectants or both. There are also bath emollients and directly applied ones. Very little has been studied regarding their effectiveness. Emollients available may also contain preservatives and fragrances that can prove to be irritants when applied topically (Rubel et al., 2013).
5. Rice bran and products derived from it have been studied regarding their anti-oxidant, nutritional, cholesterol lowering and health promoting properties (Nagendra Prasad et al., 2011).

   However, there are very few studies that have focused on the benefits of SWRB when used topically.
6. Justification: SWRB is cost-effective and easily available, while being an under-utilised product. The investigators wanted to study its effectiveness in controlling the signs and symptoms of Atopic Dermatitis when used as a cleanser and topical paste (emollient) as very little is known on this subject.

Methodology This is a clinical trial involving topical therapy with pure SWRB which is in powder form, on patients below 18 years of age, who suffer from mild to moderate atopic dermatitis. The SWRB is from locally grown rice and locally milled rice bran. This has been recently stabilised, for the first time in Malaysia, and made suitable for human use by Rice Bran Nutraceuticlas Sdn. Bhd (RBN). The SWRB is provided Free of Charge for this Study by RBN.

Sample size: The proposed sample size is 50-100 patients of the above mentioned age group.

The severity of disease in the selected sample will be assessed using the widely used SCORAD index.

Patients will be selected from out-patient clinics of

* Dato' Dr S Sellappan's clinic at Loh Guan Lye Specialist Centre.
* Klinik Derma Sivasantha at 11, Jalan Sungai. 10150 Pulau Pinang.
* Any other Doctor or Clinic who is interested in participating in this study. Written consent to participate in this study will be obtained from the parent/guardian via a consent form, which includes Information Leaflet for the Parent/Guardian and Participant as well as Instructions to Patients for Use of SWRB as cleanser or as moisturiser. Assent from the subjects from the ages from 8 to below 18 will be obtained using the assent form attached. Both, the consent and the assent forms will be attached to the child's medical records. Confidentiality of patient information and anonymity will be maintained at all times.

Proposed intervention:

Patients with mild AD will be given SWRB in powder form, to be used as a cleanser after adding water to it according to set proportions given as instructions, one time per day.

Patients with moderate disease will be instructed to use SWRB as a cleanser as above. In addition, they will also use SWRB as an emollient after constituting it into a paste as in instructions, apply at night and leave it overnight. This study does not involve any enteral or parenteral administration of SWRB.

Neither does it involve any invasive procedures.

Data collection The patients will be followed up for four to six (4 - 6) weeks and the clinical features tabulated . Where appropriate, photographs of the lesion/s will be taken for evaluation of progression / regression at the end of the study, while protecting the identity of the patient.

A questionnaire using the Likert scale, will be prepared for the patient's parent/s to complete. This will be to assess:

* Parents' opinion of the product
* Ease of application
* Convenience (cleaning the bed of the powder, etc.)
* Parents' perception regarding improvement seen/not seen

Duration of study The study will commence on 21st September 2020. The duration of this study will be 4 to 6 weeks i.e. each participant will be followed up for 4 - 6 weeks for the purpose of obtaining results for this study. However, follow up beyond the duration of this study may continue as per participants' wishes, for the purpose of continued therapy of the long -term condition, which may or may not involve SWRB. Each participant will be followed up every two (2) weeks and the progression or regression of the skin lesions recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients below 18 years of age with mild and moderate Atopic Dermatitis

Exclusion Criteria:

1. Those over 18 years of age
2. Patients with other forms of dermatitis
3. Severe disease
4. Those already on other forms of topical therapies, which are likely to interfere with outcomes

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
SCORAD index change | 0 weeks
  Used to assess the effectiveness of treatment, done before treatment. http://scorad.corti.li/
SCORAD index change | 2 weeks
  Used to assess the effectiveness of treatment, done during treatment. http://scorad.corti.li/
SCORAD index change | 4 weeks
  Used to assess the effectiveness of treatment, done after treatment. http://scorad.corti.li/

CONTACTS AND LOCATIONS:
Overall Officials: Sellappan S, Principal Investigator — Loh Guan Lye Specialist Centre 238, Jalan Macalister 10400 George Town, Penang, Malaysia
Locations (1):
- Loh Guan Lye Specialist Centre 238, Jalan Macalister 10400 George Town Pulau Pinang, George Town, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Data collection and storage will be in accordance with the data protection laws and regulations of Malaysia. All data will be stored in a password protected electronic form accessible to and managed by the Principal Investigator. The results of the study and protocol may be shared with others if published.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: If the results are published in a journal. Time frame not available.
Access Criteria: Those who subscribe to the publication

REFERENCES:
- [Background] Carroll CL, Balkrishnan R, Feldman SR, Fleischer AB Jr, Manuel JC. The burden of atopic dermatitis: impact on the patient, family, and society. Pediatr Dermatol. 2005 May-Jun;22(3):192-9. doi: 10.1111/j.1525-1470.2005.22303.x. PMID 15916563
- [Background] Chan YC, Tay YK, Sugito TL, Boediardja SA, Chau DD, Nguyen KV, Yee KC, Alias M, Hussein S, Dizon MV, Roa F, Chan YH, Wananukul S, Kullavanijaya P, Singalavanija S, Cheong WK. A study on the knowledge, attitudes and practices of Southeast Asian dermatologists in the management of atopic dermatitis. Ann Acad Med Singap. 2006 Nov;35(11):794-803. PMID 17160196
- [Background] Fujiwaki T, Furusho K. The effects of rice bran broth bathing in patients with atopic dermatitis. Acta Paediatr Jpn. 1992 Oct;34(5):505-10. doi: 10.1111/j.1442-200x.1992.tb00997.x. PMID 1442022
- [Background] Goh YY, Keshavarzi F, Chew YL. Prevalence of Atopic Dermatitis and Pattern of Drug Therapy in Malaysian Children. Dermatitis. 2018 May/Jun;29(3):151-161. doi: 10.1097/DER.0000000000000376. PMID 29762208
- [Background] Lee J, Bielory L. Complementary and alternative interventions in atopic dermatitis. Immunol Allergy Clin North Am. 2010 Aug;30(3):411-24. doi: 10.1016/j.iac.2010.06.006. PMID 20670822
- [Background] Rubel D, Thirumoorthy T, Soebaryo RW, Weng SC, Gabriel TM, Villafuerte LL, Chu CY, Dhar S, Parikh D, Wong LC, Lo KK; Asia-Pacific Consensus Group for Atopic Dermatitis. Consensus guidelines for the management of atopic dermatitis: an Asia-Pacific perspective. J Dermatol. 2013 Mar;40(3):160-71. doi: 10.1111/1346-8138.12065. Epub 2013 Jan 5. PMID 23289827

DOCUMENTS (2):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT04635072/Prot_000.pdf
  • Informed Consent Form (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT04635072/ICF_001.pdf